CLINICAL TRIAL: NCT05171166
Title: Neoadjuvant HAIC of TACE Plus Donafenib in BCLC B Stage Hepatocellular Carcinoma Out Up-to-seven: a Multi-center Randomized Controlled Trial.
Brief Title: Neoadjuvant HAIC of TACE Plus Donafenib in BCLC B Stage HCC: a Multi-center Randomized Controlled Trial.
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Difficult to enroll participants
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Wang, MD, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-TACE
Record Dates: First submitted 2021-11-24; First posted 2021-12-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; donafenib; Glucosamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HAIC-TACE-Dona Group (Experimental): 200 mg of donafenib (consisting of two 100-mg tablets) twice daily combine with hepatic arterial infusion chemotherapy that consists of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks. After 2-4 cycles of HAIC treatment, the sequential TACE therapy would be performed.
  Interventions: Procedure: HAIC; Procedure: TACE; Drug: FOLFOX; Drug: cTACE or DEB-TACE; Drug: Donafenib
- TACE-Dona Group (Active Comparator): 200 mg of donafenib (consisting of two 100-mg tablets) twice daily combine with cTACE or DEB-TACE that mixed with EPI.
  Interventions: Procedure: TACE; Drug: cTACE or DEB-TACE; Drug: Donafenib

INTERVENTIONS:
Procedure: HAIC — Hepatic arterial infusion chemotherapy is consist of oxaliplatin (35 mg/m2 for 2 hours), followed by 5-fluorouracil (600 mg/m2 for 22 hours) on day1-3 every 4 weeks. For each cycle, leucovorin calcium 200 mg/m2 would be intravenously administered for 2 hours from beginning of 5-fluorouracil infusion.
  Arms: HAIC-TACE-Dona Group
Procedure: TACE — A standard hepatic artery catheter would be introduced via the femoral artery percutaneously. Selective catheterization of the proper hepatic artery would be performed using standard diagnostic catheters and fluoroscopic guidance. In the event of multiple arterial supply, the proportion of the liver supplied by each artery would be estimated by the arteriography. After optimal positioning of the catheter, cTACE or DEB-TACE protocol would be performed to embolize the tumor supplying artery blood flow until the stasis of the supplying artery.
Drug: FOLFOX — oxaliplatin,leucovorin, and 5-FU
  Other Names: oxaliplatin; leucovorin; 5-fluorouracil
  Arms: HAIC-TACE-Dona Group
Drug: cTACE or DEB-TACE — lipiodol or microspheres that mixed with EPI
  Other Names: EPI
Drug: Donafenib — 200 mg of donafenib (consisting of two 100-mg tablets) twice daily.
  Other Names: Dona

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the combination therapy with HAIC-TACE and donafenib compared to TACE plus donafenib in patients with BCLC B stage unresectable hepatocellular carcinoma (HCC) out of up-to-seven criteria.

DETAILED DESCRIPTION:
Trans-arterial chemoembolization (TACE) is the most widely used palliative treatment for BCLC B stage hepatocellular carcinoma (HCC) patients. While a number of studies demonstrated poor effect of TACE for patients with large hepatocellular carcinoma especially for those with tumor that out of up-to-7 criteria. Some recent studies suggested that, compared with TACE, hepatic arterial infusion chemotherapy (HAIC) may improve the survivals for HCC with large tumor. Thus, the investigators carried out this prospective randomized controlled trial to demonstrate the superiority of neoadjuvant HAIC of TACE.

Total 156 subjects will be recruited in this study, each group of 78 subjects in treatment group (HAIC-TACE-Dona group) and control group (TACE-Dona group). Primary efficacy analysis will be done in the full analysis set. PFS will be used as primary outcome measures. OS, TTP, ORR, DCR and safety will be the secondary endpoints. In addition, the safety evaluation will be carried out according to the standard of adverse reaction classification (Common Terminology Criteria for Adverse Events, CTCAE v5.0).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must volunteer to participate in the study, signed informed consent, and were able to comply with the program requirements of visits and related procedures.
2. Age and gender: >18 years old and≤75 years old, both men and women.
3. All subjects must have Hepatocellular Carcinoma confirmed by pathological or clinical diagnosis.
4. Subjects are not suitable for radical resection or radical ablative therapy.
5. BCLC B based on Barcelona Clinic Liver Cancer staging system, and the lesions in the liver exceed up to 7 criteria, the number of tumors + the maximum diameter of tumors > 7.
6. Patients with viable and measurable target lesion per mRECIST.
7. Patients who are expected to live more than 3 months.
8. ECOG PS 0-1.
9. Child-Pugh class A.
10. Patients with laboratory values that meet the following criteria:

    1. Hemoglobin≥90 g/L;
    2. Neutrophile granulocytes≥1.5×109/L;
    3. Platelet count≥75×109/L;
    4. Albumin≥30 g/L;
    5. Total serum bilirubin ≤ 2 times upper limits of normal;
    6. AST and ALT ≤ 5 times upper limits of normal;
    7. Serum creatinine ≤ 1.5 times upper limits of normal;
    8. Alkaline phosphatase ≤ 5 times upper limits of normal;
    9. Prothrombin time or international normalized ratio ≤ 1.5 times upper limits of normal, activated partial thromboplastin time (APTT) ≤ 1.5×ULN;

Exclusion Criteria:

1. Fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma confirmed by histology or cytology.
2. History of malignant tumor, excluding the following cases:

   1. Malignant tumor that was curatively treated more than 5 years prior to study entry and has not recurred since then;
   2. Successful radical resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder carcinoma, preinvasive cervix carcinoma, and other preinvasive cancers.
3. Diffuse tumor lesion.
4. The lesions load in the liver exceeds 20, the number of tumors + the maximum diameter of tumors > 20.
5. Vascular invasion or extrahepatic metastasis.
6. Preexisting or history of hepatic encephalopathy, hepatorenal syndrome or liver transplantation.
7. Clinically uncontrolled ascites or pleural effusion.
8. History of surgical excision or ablation within 4 weeks of the start of treatment.
9. History of hepatic arterial infusion, more than twice TACE therapy, or history of TACE within 6 months of the start of treatment.
10. History of systemic therapy, including but not limited to chemotherapy, targeted therapy, immunotherapy.
11. History of thrombosis and/or embolism within 6 months of the start of treatment.
12. Clinically severe gastrointestinal bleeding within 6 months of the start of treatment or any life-threatening bleeding events within 3 months of the start of treatment.
13. Clinically significant cardiovascular disease, including, but not limited to, acute myocardial infarction, severe/unstable angina or prior coronary artery bypass surgery, congestive heart failure (NYHA >2), poorly controlled arrhythmias or arrhythmias requiring pacemaker therapy, hypertension not controlled by medication (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) within the past 6 months.
14. Other significant clinical and laboratory abnormalities, such as uncontrolled diabetes, chronic kidney disease, grade II or above peripheral neuropathy (CTCAE V5.0), and thyroid dysfunction, that may affect the safety evaluation.
15. Severe infections that are active or clinically poorly controlled.
16. If accompanied by acute or chronic active hepatitis B, unless taking antiviral drugs.
17. Female patients who are pregnant, lactating, possibly pregnant, or planning to become pregnant, and fertile female or male patient who is unwilling or unable to use effective contraception.
18. Multiple branches of hepatic artery with severe variation.
19. Any other subjects that the investigator considers ineligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-24 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of treatment beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  The date from the initiation of treatment to the date that disease progression or death due to any cause, whichever occurs firstly.

SECONDARY OUTCOMES:
Overall Survival | From date of treatment beginning until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.
  The date from the initiation of treatment to the date of death.
Time To Progression | Evaluation of tumor burden based on mRECIST criteria until first documented progress, assessed up to 100 months.
  Time to progression is defined as time from treatment initiation to radiological progression.
Objective response rate | Evaluation of tumor burden based on mRECIST criteria through study completion, an average of once per 3 months.
  The proportion of participants in the analysis population who have complete response (CR) or partial response (PR) determined by investigators using mRECIST criteria at any time during the study.
Disease control rate | Evaluation of tumor burden based on mRECIST criteria through study completion, an average of once per 3 months.
  The proportion of participants in the analysis population who have CR, PR or stable disease (SD) determined by investigators using mRECIST criteria at any time during the study.
Number of paitents with treatment-related adverse events | Through study completion, an average of once per 1 month.
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodong Wang, MD, Principal Investigator — Department of Interventional Therapy, Peking University Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Background] Farsad K, Nabavizadeh N, Kardosh A, Jou JH, Naugler WE, Kolbeck KJ. Combined locoregional and systemic therapy for advanced hepatocellular carcinoma: finally, the future is obscure. Ann Transl Med. 2020 Dec;8(24):1700. doi: 10.21037/atm-20-4164. No abstract available. PMID 33490212
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Llovet JM, Bruix J. Systematic review of randomized trials for unresectable hepatocellular carcinoma: Chemoembolization improves survival. Hepatology. 2003 Feb;37(2):429-42. doi: 10.1053/jhep.2003.50047. PMID 12540794
- [Background] Kokudo N, Takemura N, Hasegawa K, Takayama T, Kubo S, Shimada M, Nagano H, Hatano E, Izumi N, Kaneko S, Kudo M, Iijima H, Genda T, Tateishi R, Torimura T, Igaki H, Kobayashi S, Sakurai H, Murakami T, Watadani T, Matsuyama Y. Clinical practice guidelines for hepatocellular carcinoma: The Japan Society of Hepatology 2017 (4th JSH-HCC guidelines) 2019 update. Hepatol Res. 2019 Oct;49(10):1109-1113. doi: 10.1111/hepr.13411. Epub 2019 Sep 6. PMID 31336394
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Wang Q, Xia D, Bai W, Wang E, Sun J, Huang M, Mu W, Yin G, Li H, Zhao H, Li J, Zhang C, Zhu X, Wu J, Li J, Gong W, Li Z, Lin Z, Pan X, Shi H, Shao G, Liu J, Yang S, Zheng Y, Xu J, Song J, Wang W, Wang Z, Zhang Y, Ding R, Zhang H, Yu H, Zheng L, Gu W, You N, Wang G, Zhang S, Feng L, Liu L, Zhang P, Li X, Chen J, Xu T, Zhou W, Zeng H, Zhang Y, Huang W, Jiang W, Zhang W, Shao W, Li L, Niu J, Yuan J, Li X, Lv Y, Li K, Yin Z, Xia J, Fan D, Han G; China HCC-TACE Study Group. Development of a prognostic score for recommended TACE candidates with hepatocellular carcinoma: A multicentre observational study. J Hepatol. 2019 May;70(5):893-903. doi: 10.1016/j.jhep.2019.01.013. Epub 2019 Jan 18. PMID 30660709
- [Background] Wang Q, Xia D, Bai W, Wang E, Han G. Reply to: "The "six-and-twelve score" for TACE treatment: Does it really help us?". J Hepatol. 2019 Nov;71(5):1053-1054. doi: 10.1016/j.jhep.2019.07.009. Epub 2019 Sep 26. No abstract available. PMID 31500855
- [Background] Arizumi T, Minami T, Chishina H, Kono M, Takita M, Yada N, Hagiwara S, Minami Y, Ida H, Ueshima K, Kamata K, Minaga K, Komeda Y, Takenaka M, Sakurai T, Watanabe T, Nishida N, Kudo M. Time to Transcatheter Arterial Chemoembolization Refractoriness in Patients with Hepatocellular Carcinoma in Kinki Criteria Stages B1 and B2. Dig Dis. 2017;35(6):589-597. doi: 10.1159/000480208. Epub 2017 Oct 17. PMID 29040992
- [Background] Tsurusaki M, Murakami T. Surgical and Locoregional Therapy of HCC: TACE. Liver Cancer. 2015 Sep;4(3):165-75. doi: 10.1159/000367739. Epub 2015 Jul 10. PMID 26675172
- [Background] Golfieri R, Giampalma E, Renzulli M, Cioni R, Bargellini I, Bartolozzi C, Breatta AD, Gandini G, Nani R, Gasparini D, Cucchetti A, Bolondi L, Trevisani F; PRECISION ITALIA STUDY GROUP. Randomised controlled trial of doxorubicin-eluting beads vs conventional chemoembolisation for hepatocellular carcinoma. Br J Cancer. 2014 Jul 15;111(2):255-64. doi: 10.1038/bjc.2014.199. Epub 2014 Jun 17. PMID 24937669
- [Background] Sacco R, Bargellini I, Bertini M, Bozzi E, Romano A, Petruzzi P, Tumino E, Ginanni B, Federici G, Cioni R, Metrangolo S, Bertoni M, Bresci G, Parisi G, Altomare E, Capria A, Bartolozzi C. Conventional versus doxorubicin-eluting bead transarterial chemoembolization for hepatocellular carcinoma. J Vasc Interv Radiol. 2011 Nov;22(11):1545-52. doi: 10.1016/j.jvir.2011.07.002. Epub 2011 Aug 16. PMID 21849247
- [Background] Angelico M. TACE vs DEB-TACE: Who wins? Dig Liver Dis. 2016 Jul;48(7):796-7. doi: 10.1016/j.dld.2016.05.009. Epub 2016 May 17. No abstract available. PMID 27257050
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Kudo M, Ueshima K, Ikeda M, Torimura T, Tanabe N, Aikata H, Izumi N, Yamasaki T, Nojiri S, Hino K, Tsumura H, Kuzuya T, Isoda N, Yasui K, Aino H, Ido A, Kawabe N, Nakao K, Wada Y, Yokosuka O, Yoshimura K, Okusaka T, Furuse J, Kokudo N, Okita K, Johnson PJ, Arai Y; TACTICS study group. Randomised, multicentre prospective trial of transarterial chemoembolisation (TACE) plus sorafenib as compared with TACE alone in patients with hepatocellular carcinoma: TACTICS trial. Gut. 2020 Aug;69(8):1492-1501. doi: 10.1136/gutjnl-2019-318934. Epub 2019 Dec 4. PMID 31801872
- [Background] Qu XD, Chen CS, Wang JH, Yan ZP, Chen JM, Gong GQ, Liu QX, Luo JJ, Liu LX, Liu R, Qian S. The efficacy of TACE combined sorafenib in advanced stages hepatocellullar carcinoma. BMC Cancer. 2012 Jun 21;12:263. doi: 10.1186/1471-2407-12-263. PMID 22721173
- [Background] Wan X, Zhai X, Yan Z, Yang P, Li J, Wu D, Wang K, Xia Y, Shen F. Retrospective analysis of transarterial chemoembolization and sorafenib in Chinese patients with unresectable and recurrent hepatocellular carcinoma. Oncotarget. 2016 Dec 13;7(50):83806-83816. doi: 10.18632/oncotarget.11514. PMID 27566566
- [Background] Yao X, Yan D, Zeng H, Liu D, Li H. Concurrent sorafenib therapy extends the interval to subsequent TACE for patients with unresectable hepatocellular carcinoma. J Surg Oncol. 2016 May;113(6):672-7. doi: 10.1002/jso.24215. Epub 2016 Mar 14. PMID 26989044
- [Background] Zhong BY, Ni CF, Chen L, Zhu HD, Teng GJ. Early Sorafenib-related Biomarkers for Combination Treatment with Transarterial Chemoembolization and Sorafenib in Patients with Hepatocellular Carcinoma. Radiology. 2017 Aug;284(2):583-592. doi: 10.1148/radiol.2017161975. Epub 2017 Mar 6. PMID 28263701
- [Background] Yao Q, Zhang H, Xiong B, Zheng C. Combination of sorafenib and TACE inhibits portal vein invasion for intermediate stage HCC: a single center retrospective controlled study. Oncotarget. 2017 Sep 8;8(45):79012-79022. doi: 10.18632/oncotarget.20745. eCollection 2017 Oct 3. PMID 29108283
- [Background] Zhu K, Huang J, Lai L, Huang W, Cai M, Zhou J, Guo Y, Chen J. Medium or Large Hepatocellular Carcinoma: Sorafenib Combined with Transarterial Chemoembolization and Radiofrequency Ablation. Radiology. 2018 Jul;288(1):300-307. doi: 10.1148/radiol.2018172028. Epub 2018 Apr 24. PMID 29688153
- [Background] Lei XF, Ke Y, Bao TH, Tang HR, Wu XS, Shi ZT, Lin J, Zhang ZX, Gu H, Wang L. Effect and safety of sorafenib in patients with intermediate hepatocellular carcinoma who received transarterial chemoembolization: A retrospective comparative study. World J Clin Cases. 2018 May 16;6(5):74-83. doi: 10.12998/wjcc.v6.i5.74. PMID 29774219
- [Background] Ren B, Wang W, Shen J, Li W, Ni C, Zhu X. Transarterial Chemoembolization (TACE) Combined with Sorafenib versus TACE Alone for Unresectable Hepatocellular Carcinoma: A Propensity Score Matching Study. J Cancer. 2019 Jan 29;10(5):1189-1196. doi: 10.7150/jca.28994. eCollection 2019. PMID 30854128
- [Background] Qin S, Bi F, Gu S, Bai Y, Chen Z, Wang Z, Ying J, Lu Y, Meng Z, Pan H, Yang P, Zhang H, Chen X, Xu A, Cui C, Zhu B, Wu J, Xin X, Wang J, Shan J, Chen J, Zheng Z, Xu L, Wen X, You Z, Ren Z, Liu X, Qiu M, Wu L, Chen F. Donafenib Versus Sorafenib in First-Line Treatment of Unresectable or Metastatic Hepatocellular Carcinoma: A Randomized, Open-Label, Parallel-Controlled Phase II-III Trial. J Clin Oncol. 2021 Sep 20;39(27):3002-3011. doi: 10.1200/JCO.21.00163. Epub 2021 Jun 29. PMID 34185551